CLINICAL TRIAL: NCT05151341
Title: Evaluation of a Urine Analysis Combining VisioCyt® Automated Cytology and FGFR3 Mutations for the Detection of Bladder Cancer
Brief Title: Study of Combined VisioCyt Test and FGFR3 Mutations on a Urinary Sample to Diagnose Bladder Tumors
Acronym: URODX-FGFR3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Collaborators: Vitadx (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-A01054-37
Record Dates: First submitted 2021-12-01; First posted 2021-12-09 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2024-12

CONDITIONS: Bladder Cancer
Keywords: FGFR3; VisioCyt; Bladder Tumor; Cancer; FGFR3 Mutation; Diagnosis; Cytoloogy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplasms; Disease | interventions — Urine Specimen Collection; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Case (Experimental): Patient in whom newly diagnosed, or recurring / progressing bladder cancer is strongly suspected after initial fibroscopy
  Interventions: Diagnostic Test: Urine collection (150ml); Other: Blood sample (20 ml)
- Control (Experimental): Patient attending or hospitalized for urolithiasis, urinary infections, superior excretory stones or with non suspect urinary symptomatology
  Interventions: Diagnostic Test: Urine collection (150ml)

INTERVENTIONS:
Diagnostic Test: Urine collection (150ml) — Urine collection will be tacken at inclusion. The sample will be thereafter separate into three to realise different analyzes (standard cytology, Visiocyt test, FGFR3 analysis)
Other: Blood sample (20 ml) — Blood sample will be tacken at inclusion, ONLY for "case" patients that agreed upon this. This sample will be addition to the collection for further research.
  Arms: Case

SUMMARY:
This study is a case-control, propsective and muticentric clinical trial, which aim to compare the specificity and sensibility of VisioCyt urinary cytological test combined with FGFR3 mutation detection test to VisioCyt urinary cyological test on its own to detect bladder cancer.

The case are patient in whom newly diagnosed, or recurring /progressing bladder cancer is strongly suspected after initial fibroscopy.

The control are patient attending or hospitalized for urolithiasis, urinary infections, urinary superior excretory stones or with non suspect urinary symptomatology.

ELIGIBILITY:
INCLUSION CRITERIA

BOTH GROUPS

* M/F
* Patient agrees to follow study protocol and is able to follow study procedures
* Patient signed, dated and understood consent form
* Patient has a social security scheme

CASE GROUP

* Patient is 18 or older
* Patient for whom a bladder cancer recently diagnosed, or backsliding/progression is heavily suspected after the initial fibroscopy
* Patient who hasn't started systemic/oral/radiotheurapeutic pelvic treatment for his/her tumor

CONTROL GROUP

* Patient between 18 and 45 y/o
* Patient not suspected of having any bladder cancer
* Patient attending or hospitalized for urolithiasis, urinary infections, superior excretory stones or with non suspect urinary symptomatology
* Patient who hasn't been exposed to bladder carcinogens (tobacco, industrial carcinogen (ex: coal tar, tar/coal oils, coal pitch and burning coal soot), urinary bilharzia, chemotherapy exposition (cyclophosphamid)
* Patient that had a negative cytopathological exploration of the excretory urinary route OR/AND iconography (pelvic echography, pelvic scanner) OR/AND endoscopy with prior urinary sample
* Patient unscathed of any cancer that might interact with bladder cancer : uterine cancer, prostate cancer, rectal cancer, and metastasis from other cancer or non-urologic tumor invading the bladder

EXCLUSION CRITERIA BOTH GROUPS

* Non-treated current urinary infection
* Patient with another pelvic cancer
* Bladder cancer outside of urothelial carcinoma
* Associated carcinoma of the high urinary apparatus
* Patient that received renal transplantation (BK virus)
* Patient that received pelvis radiotherapy (related to prostatic cancer, gynecologic cancer or pelvic digestive cancer)
* Patient having a JJ catheter
* Refused to signed consent
* Pregnant, susceptible to be, or breast-feeding women
* Person Under guardianship
* Impossibility to submit to medical monitoring because of geographic, social, or mental issues

CASE GROUP • Under 18y/o

CONTROL GROUP

• Under 18y/o or above 45 y/o

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Specificity | at inclusion
  Specificity comparaison between Visiocyt test + FGFR3 analysis and FGFR3 analysis on its own

SECONDARY OUTCOMES:
Sensitivity of the 4 different tests | at inclusion
  Sensibility Comparaison between :
  1. Visiocyt test + FGFR3 analysis
  2. FGFR3 analysis on its own
  3. Visiocyt test on its own
  4. Standard cytology
Specificity of the 4 different tests | at inclusion
  Specificity Comparaison between :
  1. Visiocyt test + FGFR3 analysis
  2. FGFR3 analysis on its own
  3. Visiocyt test on its own
  4. Standard cytology
Positive predictive value of the 4 different tests | at inclusion
  Positive predictive value between :
  1. Visiocyt test + FGFR3 analysis
  2. FGFR3 analysis on its own
  3. Visiocyt test on its own
  4. Standard cytology
Negative predictive value of the 4 different tests | at inclusion
  Negative predictive value between :
  1. Visiocyt test + FGFR3 analysis
  2. FGFR3 analysis on its own
  3. Visiocyt test on its own
  4. Standard cytology

CONTACTS AND LOCATIONS:
Overall Officials: Eschwège Pascal, MD, PhD, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, France